CLINICAL TRIAL: NCT04785261
Title: Pilot Study on The Effect of Traditional Chinese Medicine on Basic Tear Secretion and Tear Cytokines in Patients With Dry Eye Disease
Brief Title: Effect of Traditional Chinese Medicine on Basic Tear Secretion and Tear Cytokines in Patients With Dry Eye Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH109-REC2-169
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Disease; Dry Eye Syndromes; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — carbomer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Active Comparator): Patients in this group will be given conventional treatment including Artelac® Eye Drops (1-2 drips each time, every 4 hours) and Vidisic® Gel (1 drip each time, at bedtime) for 12 weeks.
  Interventions: Drug: Methylhydroxypropylcellulose; Drug: Carbomer
- conventional treatment + TCM (Experimental): Patients in this group will be given conventional treatment and traditional Chinese medicine (6.0g twice daily) for 12 weeks.
  Interventions: Drug: Methylhydroxypropylcellulose; Drug: Carbomer; Drug: TCM Formula

INTERVENTIONS:
Drug: Methylhydroxypropylcellulose — 1-2 drips each time, every 4 hours, for 12 weeks.
  Other Names: Artelac® Eye Drops
Drug: Carbomer — 1 drip each time, at bedtime, for 12 weeks.
  Other Names: Vidisic® Gel
Drug: TCM Formula — 6.0g Chi-Ju-Di-Huang-Wan plus 6.0g Jia-Wei-Xiao-Yao-San, 6.0g twice daily for 12 weeks.
  Arms: conventional treatment + TCM

SUMMARY:
This is a single center, randomized, single-blind, controlled pilot study of CJDHW plus JWXYS as a complementary therapy to treat dry eye disease during a 12-week period. The investigators intend to enroll 60 subjects aged between 20 and 75 years old (treatment group(N=30); controlled group(N=30)). Treatment group will be treated with artificial tears combined with TCM, while control group will use artificial tears only. The aim of this study is to explore the efficacy of TCM for dry eye disease.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a chronic inflammatory disease. In severe cases, it may cause corneal ulcers, blurred vision, and even blindness. The prevalence of DED is about 30% in Taiwan. With the popularity of technological products and prolonged average life expectancy, the incidence of dry eye disease is increasing at a rate of 10% per year in Taiwan. However, treatment of DED mainly focuses on symptom relief in modern medicine. It is a difficult problem to improve the pathological state of patients with DED. Hence, there is an urgent need for a more effective and safe method of treating this disease.

Chi-Ju-Di-Huang-Wan (CJDHW) is commonly used in traditional Chinese medicine (TCM) for eye diseases. However, current research shows that use CJDHW alone to treat dry eye is less effective for tear secretion, which may be related to the unimproved inflammation state. Ligustilide and ferulic acid, which own significant anti-inflammatory effects, are the effective ingredients of Jia-Wei-Xiao-Yao-San (JWXYS). Many studies have demonstrated that JWXYS can reduce serum TNF-α and IFN-γ levels in patients with DED. Therefore, the investigators choose to use CJDHW plus JWXYS for treatment in this study.

This is a single center, randomized, single-blind, controlled pilot study of CJDHW plus JWXYS as a complementary therapy to treat dry eye disease during a 12-week period. The investigators intend to enroll 60 subjects aged between 20 and 75 years old (treatment group(N=30); controlled group(N=30)). Treatment group will be treated with artificial tears combined with TCM, while control group will use artificial tears only. The evaluation will be conducted on 1st, 4th, 8th,12th week. Primary endpoints include Schirmer's test and non-invasive tear film breakup time(NiBUT); secondary endpoints include tear meniscus height, meibomian gland loss rate, tear cytokines and matrix metalloproteinases (MMPs) levels and Ocular Surface Disease Index (OSDI).

The aim of this study is to explore the efficacy and possible mechanism of TCM for DED.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 75 years.
* A confirmed diagnosis of DED by ophthalmologists.
* Willing to sign informed consent form.

Exclusion Criteria:

* With autoimmune diseases.
* Pregnant or lactating.
* Underwent transplant surgery and got graft-versus-host disease in the past.
* With eye infection, inflammation, trauma, or underwent eye surgery in the past three months.
* Underwent dry eye intense pulse light treatment in the past three months.
* Underwent other treatments including TCM drugs or acupuncture in the past month or during the trial.
* Persistent in taking diuretics, antidepressant, antihistamines and anticholinergics.
* Combined treatment with autologous serum, cyclosporine or steroid eye drops during the trial.
* Took fish oil or vitamin D during the trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Schirmer's Test | Change from baseline Schirmer's Test at week 4, week 8 and week 12
  Uses paper strips inserted into the eye for 5 minutes to measure the production of tears. Both eyes are tested at the same time.
Non-invasive Tear Film Break-up Time (NiBUT) | Change from baseline NiBUT at week 4, week 8 and week 12
  Measured by Antares Corneal Topography.

SECONDARY OUTCOMES:
Tear Meniscus Height | Change from baseline Tear meniscus height at week 4, week 8 and week 12
  Measured by Antares Corneal Topography.
Meibomian Gland Loss Rate | Change from baseline Meibomian gland loss rate at week 4, week 8 and week 12
  Measured by Antares Corneal Topography.
Tear Cytokines | Change from baseline Tear cytokines at week 4, week 8 and week 12
Ocular Surface Disease Index (OSDI) | Change from baseline OSDI at week 4, week 8 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Lin, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan